CLINICAL TRIAL: NCT02956070
Title: Evaluation of Anti-inflammatory Steroids of Use in the Prevention of Tooth Sensitivity in Teeth Whitening Technique Office
Brief Title: Anti-inflammatory Steroids in the Prevention of Tooth Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal Fluminense (Other)
Responsible Party: Principal Investigator, Luiz Augusto da Costa Poubel, Professor, Universidade Federal Fluminense
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: bleaching
Record Dates: First submitted 2016-10-25; First posted 2016-11-04 (Estimated); Results first posted 2020-11-25 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: Inflammation
Keywords: dental bleaching; antiinflammatory; tooth sensitivity
MeSH Terms: conditions — Inflammation; Dentin Sensitivity | interventions — dexamethasone acetate; Dexamethasone; potassium nitrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): 35 patients in this group will undergo the whitening procedure using the Dexamethasone acetate intervention.
  Interventions: Drug: Dexamethasone acetate
- Placebo (Placebo Comparator): 35 patients in this group will undergo the whitening procedure using the Potassium Nitrate intervention
  Interventions: Drug: Potassium Nitrate

INTERVENTIONS:
Drug: Dexamethasone acetate — The volunteers in the Dexamethasone acetate group (experimental group) will receive six capsules of dexamethasone 8 mg each to be administered orally, initially two days before the first bleaching query as follows: 8 mg (1 capsule) 9 am two days before the first clinical session whitening; 8 mg (1 capsule) the 9 am to 1 day before session whitening, 8 mg (1 capsule) to 9 am on the day of the first session of whitening.Clinical intervention: 1- Dry teeth and apply Gingival Barrier to both arches. 2- Light cure. 3- Firmly attach a mixing nozzle to the Pola Office+. 4- Apply a thin layer of gel to all teeth undergoing treatment. 5- Leave gel on for 8 minutes. 6- Suction it off. 7- Repeat steps 5-6 twice times. 8- After the last application, suction all the gel off, then wash and apply suction. 9- Remove Gingival Barrier. 10- A placebo gel will be applied with a brush on the labial surface of the teeth whitened for 2 to 3 minutes .
  Other Names: Dexamethasone
  Arms: Experimental
Drug: Potassium Nitrate — The volunteers in the Potassium Nitrate Group (Placebo group) will receive 6 placebo capsules, who contained the same components of de dexamethasone drug except the active ingredient (starch [50%], lactose monohydrate [35%], dibasic calcium phosphate [14%], and magnesium stearate [1%]).Clinical session:1- Dry teeth and apply Gingival Barrier to both arches. 2- Light cure. 3- Firmly attach a mixing nozzle to the Pola Office+. 4- Apply a thin layer of gel to all teeth undergoing treatment. 5- Leave gel on for 8 minutes. 6- Suction it off. 7- Repeat steps 5-6 twice times. 8- After the last application, suction all the gel off, then wash and apply suction. 9- Remove Gingival Barrier. 10- A desensitizing gel containing 6% potassium nitrate will be applied with a brush on the labial surface of the teeth whitened for 2 to 3 minutes .
  Other Names: Smoothe SDI
  Arms: Placebo

SUMMARY:
Clinical randomized, triple-blind, used to measure the level of tooth sensitivity on volunteers using a modified virtual analog scale (VAS). Sixty-six volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion. All volunteers will be guided and sign a term of clarification and consent. Volunteers will be randomly divided into two groups: the control group to receive placebo capsules and application of desensitizing gel containing 6% potassium nitrate and 0.10% fluoro- (conventional treatment) and the experimental group will receive the anti-inflammatory corticosteroids (dexamethasone, capsule - 8mg) and application of a placebo gel. Patients will be treated in two clinical sessions with an interval of 7 days (one week) between them. The protocol for use of the product is as follows: The volunteers in the experimental group will receive six capsules of dexamethasone 8 mg each to be administered orally, initially two days before the first bleaching query as follows: 8 mg (1 capsule) 9 am in the morning two days before the first clinical session whitening; 8 mg (1 capsule) the 9 am to 1 day before the first practice session whitening, 8 mg (1 capsule) to 9 am on the day of the first practice session of whitening. After 7 days (one week), the same protocol will be held for the second and final practice session office bleaching.

DETAILED DESCRIPTION:
The experimental design will follow the consolidated standards for test reports (CONSORT). After approval by the Ethics Committee for Research duly registered, the trial will be conducted in the clinic of dental school at the Federal Fluminense University located in Nova Friburgo.Every Health Institute participants will be informed about the nature and objectives of the study.It will be one test study Clinical randomized, parallel, triple-blind, used to measure the level of tooth sensitivity volunteers using a modified virtual analog scale (VAS). Sixty-six volunteers will be selected and recruited, following inclusion criteria and pre-established exclusion. All volunteers will be guided and sign a term of clarification and consent. Volunteers will be randomly divided into two groups: the control group to receive placebo capsules and application of desensitizing gel containing 6% potassium nitrate and 0.10% fluoro- (conventional treatment) and the experimental group will receive the anti-inflammatory corticosteroids (dexamethasone, capsule - 8mg) and application of a placebo gel. Patients will be treated in two clinical sessions with an interval of 7 days (one week) between them. The protocol for use of the product is as follows: The volunteers in the experimental group will receive six capsules of dexamethasone 8 mg each to be administered orally, initially two days before the first bleaching query as follows: 8 mg (1 capsule) 9 am in the morning two days before the first clinical session whitening; 8 mg (1 capsule) the 9 am to 1 day before the first practice session whitening, 8 mg (1 capsule) to 9 am on the day of the first practice session of whitening. After 7 days (one week), the same protocol will be held for the second and final practice session office bleaching.

ELIGIBILITY:
Inclusion Criteria:

* The selected volunteers should present a good general state of health, be at least 18 years of age, regardless of gender, color / race and ethnicity, sexual orientation, and gender identity.
* Volunteers must have an acceptable oral hygiene, present the upper and lower arches without absence of teeth of first premolar right to the left first premolar.
* These elements have to be healthy, that is, not having any kind of restoration.
* Volunteers must sign the consent form and clarification, have committed to return for periodic examinations and belong to the group of nonsmokers.

Exclusion Criteria:

* Do not have medical history of diseases that can affect the results of the study;
* subjects could not have made use of cigarettes in the last 30 days; have some important pathology in the oral cavity;
* not being pregnant and also are not breastfeeding;
* having any history of sensitivity or adverse reactions to anti-inflammatory used in the study;
* not having calculations or advanced periodontal disease;
* have not consumed drugs, alcohol or any medication that can cover the results, as other types of anti-inflammatories or painkillers;
* The volunteers should not have used products indicated for dental sensitivity, as desensitizing toothpaste or similar product and not present recession or exacerbated hypersensitivity history.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2015-10; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcos O Barceleiro, MSD, PhD, Principal Investigator — Fluminense Federal University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carey CM. Tooth whitening: what we now know. J Evid Based Dent Pract. 2014 Jun;14 Suppl:70-6. doi: 10.1016/j.jebdp.2014.02.006. Epub 2014 Feb 13. PMID 24929591
- [Background] de Paula EA, Loguercio AD, Fernandes D, Kossatz S, Reis A. Perioperative use of an anti-inflammatory drug on tooth sensitivity caused by in-office bleaching: a randomized, triple-blind clinical trial. Clin Oral Investig. 2013 Dec;17(9):2091-7. doi: 10.1007/s00784-013-0918-2. Epub 2013 Jan 31. PMID 23371755
- [Background] de Paula EA, Kossatz S, Fernandes D, Loguercio AD, Reis A. Administration of ascorbic acid to prevent bleaching-induced tooth sensitivity: a randomized triple-blind clinical trial. Oper Dent. 2014 Mar-Apr;39(2):128-35. doi: 10.2341/12-483-C. Epub 2013 Jun 26. PMID 23802640
- [Background] de Paula EA, Nava JA, Rosso C, Benazzi CM, Fernandes KT, Kossatz S, Loguercio AD, Reis A. In-office bleaching with a two- and seven-day intervals between clinical sessions: A randomized clinical trial on tooth sensitivity. J Dent. 2015 Apr;43(4):424-9. doi: 10.1016/j.jdent.2014.09.009. Epub 2014 Sep 23. PMID 25257824
- [Background] Bonafe E, Loguercio AD, Reis A, Kossatz S. Effectiveness of a desensitizing agent before in-office tooth bleaching in restored teeth. Clin Oral Investig. 2014 Apr;18(3):839-45. doi: 10.1007/s00784-013-1055-7. PMID 23959376
- [Background] Bonafe E, Bacovis CL, Iensen S, Loguercio AD, Reis A, Kossatz S. Tooth sensitivity and efficacy of in-office bleaching in restored teeth. J Dent. 2013 Apr;41(4):363-9. doi: 10.1016/j.jdent.2013.01.007. Epub 2013 Jan 26. PMID 23357647
- [Background] Faria-E-Silva AL, Nahsan FP, Fernandes MT, Martins-Filho PR. Effect of preventive use of nonsteroidal anti-inflammatory drugs on sensitivity after dental bleaching: a systematic review and meta-analysis. J Am Dent Assoc. 2015 Feb;146(2):87-93.e1. doi: 10.1016/j.adaj.2014.10.007. PMID 25637206
- [Background] He LB, Shao MY, Tan K, Xu X, Li JY. The effects of light on bleaching and tooth sensitivity during in-office vital bleaching: a systematic review and meta-analysis. J Dent. 2012 Aug;40(8):644-53. doi: 10.1016/j.jdent.2012.04.010. Epub 2012 Apr 21. PMID 22525016
- [Background] Vadivelu N, Mitra S, Schermer E, Kodumudi V, Kaye AD, Urman RD. Preventive analgesia for postoperative pain control: a broader concept. Local Reg Anesth. 2014 May 29;7:17-22. doi: 10.2147/LRA.S62160. eCollection 2014. PMID 24872720
- [Background] Li Y, Greenwall L. Safety issues of tooth whitening using peroxide-based materials. Br Dent J. 2013 Jul;215(1):29-34. doi: 10.1038/sj.bdj.2013.629. PMID 23846062
- [Background] Markowitz K. Pretty painful: why does tooth bleaching hurt? Med Hypotheses. 2010 May;74(5):835-40. doi: 10.1016/j.mehy.2009.11.044. Epub 2009 Dec 31. PMID 20045265
- [Background] Costa CA, Riehl H, Kina JF, Sacono NT, Hebling J. Human pulp responses to in-office tooth bleaching. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2010 Apr;109(4):e59-64. doi: 10.1016/j.tripleo.2009.12.002. PMID 20303048
- [Background] Rhen T, Cidlowski JA. Antiinflammatory action of glucocorticoids--new mechanisms for old drugs. N Engl J Med. 2005 Oct 20;353(16):1711-23. doi: 10.1056/NEJMra050541. No abstract available. PMID 16236742
- [Background] Bamgbose BO, Akinwande JA, Adeyemo WL, Ladeinde AL, Arotiba GT, Ogunlewe MO. Effects of co-administered dexamethasone and diclofenac potassium on pain, swelling and trismus following third molar surgery. Head Face Med. 2005 Nov 7;1:11. doi: 10.1186/1746-160X-1-11. PMID 16274480
- [Background] Paula E, Kossatz S, Fernandes D, Loguercio A, Reis A. The effect of perioperative ibuprofen use on tooth sensitivity caused by in-office bleaching. Oper Dent. 2013 Nov-Dec;38(6):601-8. doi: 10.2341/12-107-C. Epub 2013 Apr 15. PMID 23586657
- [Background] Reis A, Tay LY, Herrera DR, Kossatz S, Loguercio AD. Clinical effects of prolonged application time of an in-office bleaching gel. Oper Dent. 2011 Nov-Dec;36(6):590-6. doi: 10.2341/10-173-C. Epub 2011 Sep 13. PMID 21913864
- [Background] Charakorn P, Cabanilla LL, Wagner WC, Foong WC, Shaheen J, Pregitzer R, Schneider D. The effect of preoperative ibuprofen on tooth sensitivity caused by in-office bleaching. Oper Dent. 2009 Mar-Apr;34(2):131-5. doi: 10.2341/08-33. PMID 19363967
- [Background] Rezende M, Bonafe E, Vochikovski L, Farago PV, Loguercio AD, Reis A, Kossatz S. Pre- and postoperative dexamethasone does not reduce bleaching-induced tooth sensitivity: A randomized, triple-masked clinical trial. J Am Dent Assoc. 2016 Jan;147(1):41-9. doi: 10.1016/j.adaj.2015.07.003. Epub 2015 Nov 6. PMID 26562735
- [Derived] da Costa Poubel LA, de Gouvea CVD, Calazans FS, Dip EC, Alves WV, Marins SS, Barcelos R, Barceleiro MO. Pre-operative use of dexamethasone does not reduce incidence or intensity of bleaching-induced tooth sensitivity. A triple-blind, parallel-design, randomized clinical trial. Clin Oral Investig. 2019 Jan;23(1):435-444. doi: 10.1007/s00784-018-2452-8. Epub 2018 Apr 25. PMID 29696420

RESULTS

PARTICIPANT FLOW:
Groups:
- Experimental: 35 patients in this group underwent the whitening procedure using the Dexamethasone acetate intervention.
  Dexamethasone acetate: The volunteers in the Dexamethasone acetate group (experimental group) received six capsules of dexamethasone 8 mg each to be administered orally, initially two days before the first bleaching query as follows: 8 mg (1 capsule) 9 am two days before the first clinical session whitening; 8 mg (1 capsule) the 9 am to 1 day before session whitening, 8 mg (1 capsule) to 9 am on the day of the first session of whitening.Clinical intervention: 1- Dry teeth and apply Gingival Barrier to both arches. 2- Light cure. 3- Firmly attach a mixing nozzle to the Pola Office+. 4- Apply a thin layer of gel to all teeth undergoing treatment. 5- Leave gel on for 8 minutes. 6- Suction it off. 7- Repeat steps 5-6 twice times. 8- After the last application, suction all the gel off, then wash and apply suction. 9- Remove Gingival Barrier. 10- A placebo gel will be applied w
- Placebo: 35 patients in this group underwent the whitening procedure using the Potassium Nitrate intervention
  Potassium Nitrate: The volunteers in the Potassium Nitrate Group (Placebo group) received 6 placebo capsules, who contained the same components of de dexamethasone drug except the active ingredient (starch [50%], lactose monohydrate [35%], dibasic calcium phosphate [14%], and magnesium stearate [1%]).Clinical session:1- Dry teeth and apply Gingival Barrier to both arches. 2- Light cure. 3- Firmly attach a mixing nozzle to the Pola Office+. 4- Apply a thin layer of gel to all teeth undergoing treatment. 5- Leave gel on for 8 minutes. 6- Suction it off. 7- Repeat steps 5-6 twice times. 8- After the last application, suction all the gel off, then wash and apply suction. 9- Remove Gingival Barrier. 10- A desensitizing gel containing 6% potassium nitrate will be applied with a brush on the labial surface of the teeth whitened for 2 to 3 minutes .
Period: Overall Study
Arm/Group | Experimental | Placebo
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Experimental: 35 patients in this group underwent the whitening procedure using the Dexamethasone acetate intervention.
  Dexamethasone acetate: The volunteers in this group received 6 capsules of dexamethasone 8 mg each to be administered orally, initially two days before the first bleaching query as follows: 8 mg (1 capsule) 9 am two days before the first clinical session whitening; 8 mg 9 am to 1 day before session whitening, 8 mg 9 am on the day of the first session of whitening.Clinical intervention: 1- Dry teeth and apply Gingival Barrier to both arches. 2- Light cure. 3- Firmly attach a mixing nozzle to the Pola Office+. 4- Apply a thin layer of gel to all teeth undergoing treatment. 5- Leave gel on for 8 minutes. 6- Suction it off. 7- Repeat steps 5-6 twice times. 8- After the last application, suction all the gel off, then wash and apply suction. 9- Remove Gingival Barrier. 10- A placebo was applied with a brush on the labial surface of the teeth whitened for 2 to 3 minutes .
- Total: Total of all reporting groups
Arm/Group | Experimental | Placebo | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.3 (2.7) | 22.5 (2.1) | 22.4 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 8 | 12 | 20
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 35 | 35 | 70

OUTCOME MEASURES:

1. Primary Outcome: Visual Analogic Scale (0-100) for Tooth Sensibility.
Description: The investigators evaluated the tooth sensibility 1 hour post-bleaching. Scale from 0-100 0 means no sensibility 100 means maximum sensibility
Time Frame: One hour
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | 6.31 (12.78) | 11.14 (20.08)

2. Primary Outcome: Visual Analogic Scale(0-100) for Tooth Sensibility.
Description: The investigators evaluated the tooth sensibility 24 hours post-bleaching. Scale from 0-100 0 means no sensibility 100 means maximum sensibility
Time Frame: Twenty four hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | 5.06 (9.86) | 8.26 (13.48)

3. Primary Outcome: Visual Analogic Scale(0-100) for Tooth Sensibility.
Description: The investigators evaluated the tooth sensibility 48 hours post-bleaching. Scale from 0-100 0 means no sensibility 100 means maximum sensibility
Time Frame: Forty eight hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Experimental | Placebo
Number analyzed (Participants) | 35 | 35
units on a scale | 0.37 (1.54) | 2.91 (9.14)

ADVERSE EVENTS:
Arm/Group | Experimental | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 0/35 | 0/35

LIMITATIONS AND CAVEATS:
No discontinuity in both treatment groups was found in the clinical investigation. All volunteers attended the recall visit 1 week postbleaching.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-20): https://cdn.clinicaltrials.gov/large-docs/70/NCT02956070/Prot_SAP_000.pdf